CLINICAL TRIAL: NCT04347980
Title: Dexamethasone Combined With Hydroxychloroquine Compared to Hydroxychloroquine Alone for Treatment of Severe Acute Respiratory Distress Syndrome Induced by Coronavirus Disease 19 (COVID-19): a Multicentre, Randomised Controlled Trial
Brief Title: Dexamethasone Treatment for Severe Acute Respiratory Distress Syndrome Induced by COVID-19
Acronym: DHYSCO
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: ANSM RECOMMANDATION
Sponsor: Centre Chirurgical Marie Lannelongue (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2037815010
Record Dates: First submitted 2020-04-09; First posted 2020-04-15 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Respiratory Distress Syndrome, Adult; COVID-19
Keywords: Acute Respiratory Distress Syndrome; COVID-19; Dexamethasone; Hydroxychloroquine; Mortality
MeSH Terms: conditions — Respiratory Distress Syndrome; COVID-19 | interventions — Dexamethasone; Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexamethasone and Hydroxychloroquine (HCQ/DXM) (Experimental): Patients included in the "HCQ / DXM" group will benefit from standardized ventilatory management and administration of HCQ in the same manner as the "HCQ" group. They will receive in addition to DXM at a rate of 20 mg intravenously for 15 min once a day for 5 days (D1 to D5) then at a rate of 10 mg per day from D6 to D10. If the patient is extubated before the 10th day, he will receive his last dose of DXM before.
  Interventions: Drug: Dexamethasone and Hydroxychloroquine
- Hydroxychloroquine (HCQ) (Active Comparator): Patients included in the "HCQ " group will benefit from standardized ventilatory management. Patients included in the "HCQ" group will receive 200 mg x 3 / day enterally from J1 of the HCQ for 10 days. If the patient is extubated before the 10th day, he will receive his last dose of HCQ before.
  Interventions: Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Dexamethasone and Hydroxychloroquine — Patients included in the "Hydroxychloroquine / Dexamethasone" group will benefit from standardized ventilatory management and administration of Hydroxychloroquine in the same manner as the Hydroxychloroquine group. They will receive in addition to Dexamethasone at a rate of 20 mg intravenously for 15 min once a day for 5 days (D1 to D5) then at a rate of 10 mg per day from D6 to D10. If the patient is extubated before the 10th day, he will receive his last dose of Dexamethasone before.
  Other Names: Standard ventilatory management
  Arms: Dexamethasone and Hydroxychloroquine (HCQ/DXM)
Drug: Hydroxychloroquine — Patients included in the Hydroxychloroquine group will benefit from standardized ventilatory management. Patients included in the Hydroxychloroquine group will receive 200 mg x 3 / day enterally from J1 of the HCQ for 10 days. If the patient is extubated before the 10th day, he will receive his last dose of HCQ before.
  Other Names: Standard ventilatory management
  Arms: Hydroxychloroquine (HCQ)

SUMMARY:
Single blind randomized clinical trial designed to evaluate the efficacy of the combination of hydroxychloroquine and dexamethasone as treatment for severe Acute Respiratory Distress Syndrome (ARDS) related to coronavirus disease 19 (COVID-19). We hypothesize that dexamethasone (20 mg for 5 days followed by 10 mg for 5 days) combined with 600 mg per day dose of hydroxychloroquine for 10 days will reduce the 28-day mortality compared to hydroxychloroquine alone in patients with severe ARDS related COVID-19.

DETAILED DESCRIPTION:
The severe acute respiratory syndrome coronavirus 2 pandemic causing COVID-19 disease affects hundreds of thousands of patients. Of these, 5% will present with acute respiratory failure, the most severe form of which is Acute Respiratory Distress Syndrome (ARDS). Hospital mortality affects 45% of patients with severe ARDS. The improvement in mortality associated with ARDS seems largely explained by the reduction in lesions induced by mechanical ventilation, in particular a tidal volume (Vt) set at 6 ml / kg of the weight predicted by the size associated with a plateau pressure must not exceed 30 cm of water. Unfortunately and despite the application of these recommendations, ARDS related COVID-19 is associated with a mortality of 65%. About 42% of patients hospitalized for COVID-19 pneumonitis will develop ARDS and the onset of ARDS is rapid after admission with a median of 2 days. Interestingly, a study reported that patients suffering from ARDS and having received corticosteroids had a mortality rate of 46% (23 out of 50) compared to 61.8% (21 out of 34) in patients who did not receive corticosteroids. However, this difference was not significant (P = 0.15). The survival curve showed, however, that the administration of corticosteroids (Methylprednisolone) reduced the risk of death (Hazard ratio: 0.38 (95% confidence interval 0.20-0.72); P = 0.003). The authors concluded that a randomized study was necessary to confirm this impression.

The theoretical justification for treatment with corticosteroids is related to the recognition of the inflammatory syndrome as a factor in the development of an uncontrolled and harmful fibroproliferative phase. It seems certain that late administration (beyond the 14th day after the start of ARDS) is deleterious in patients by increasing mortality. However, a recent study shows that early administration of dexamethasone (within 30 hours after the start of ARDS) is associated with an increase of ventilator-free days and a decrease in mortality at 2 months.

In COVID-19 disease, there is also a cytokine storm and an intense inflammatory reaction. Currently the use of corticosteroids is not recommended during a severe acute respiratory syndrome coronavirus 2 infection. Administration of corticosteroids may delay elimination of the virus. Recently, a preliminary study reported that the administration of hydroxychloroquine (200mg x3 per day) decreased or even made disappear the viral load. This clinical study appears to corroborate an experimental study. However, hydroxychloroquine can have cardiac toxicity which, although rare, can be serious.

In summary:

* The appearance of an ARDS during a COVID-19 is burdened with a mortality of 65%
* The viral load has decreased when ARDS is present
* The use of hydroxychloroquine makes it possible to significantly reduce the viral load
* Early administration of corticosteroids seems beneficial in ARDS

ELIGIBILITY:
Inclusion Criteria:

1. Patient over 18 years old
2. Patient affiliated to a health insurance plan
3. Patient who has given their free, informed and written consent or patient for whom an independent doctor has given their signed consent as part of an emergency procedure
4. Kaliemia > 3,5 mmol / L
5. Patient diagnosed COVID-19 positive by reverse transcription-polymerase chain reaction (RT-PCR) and / or CT

The diagnosis of COVID-19 will be made if:

* Patient with radiological images strongly suggestive of a chest scan associated with respiratory symptoms, without other obvious etiologies OR
* Patient with suggestive respiratory symptoms associated with a positive RT-PCR

Patients admitted to intensive care with acute respiratory distress syndrome secondary to COVID-19, intubated for less than 5 days with:

* Either - Hypoxemia defined by a arterial partial pressure of oxygen / fraction of inspiratory oxygen ratio (PaO2 / FiO2) ratio <100 after 2 sessions of prone position
* Either - An alteration in pulmonary compliance (tidal volume divided by plateau pressure minus positive expiratory pressure) immediately or over the first 96 hours after the start of ARDS defined by:
* immediately: impossibility of maintaining a plateau pressure <30 cm of water in a ventilated patient with a tidal volume of 6 ml / kg of weight predicted by the size and a positive expiratory pressure at 10 cm of water
* during the course of the evolution: decrease in compliance by 20% compared to the initial compliance (day of treatment of the intubated and ventilated patient) We define the start date of ARDS by the day and time when the patient is intubated and ventilated with regard to our definition of COVID-19

Exclusion Criteria:

1. Patient under guardianship or curator
2. Patient with plausible alternate diagnosis
3. ARDS evolving for more than 4 days
4. Contraindication to the Hydroxychloroquine : Known allergy or intolerance to the Hydroxychloroquine or to one of the excipients of the drug, in particular to lactose; documented QT prolongation and / or known risk factors for QT prolongation (including ongoing treatment with citalopram, escitalopram, hydroxyzine, domperidone or piperaquine), retinopathies
5. Contraindication to Dexamethasone: Known allergy or intolerance to Dexamethasone or to one of the excipients of the drug, another evolving virosis (hepatitis, herpes, chickenpox, shingles), severe coagulation disorder
6. Uncontrolled septic shock
7. Untreated active infection or treated less than 24 hours
8. Long-term patient treated with corticosteroids (> 20 mg / day) or Hydroxychloroquine
9. Immunocompromised patients: AIDS, bone marrow or solid organ transplant recipients
10. Pregnant women
11. Glucose-6-phosphate dehydrogenase (G6PD) deficiency

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-04-17 (Actual); Primary Completion 2020-08-07 (Actual); Study Completion 2020-08-07 (Actual)

PRIMARY OUTCOMES:
Day-28 mortality | 28 days after randomization
  Mortality rate evaluated 28 days after randomization

SECONDARY OUTCOMES:
Ventilator-free days | 28 days after randomization
  Ventilator-free days (VFDs) at 28 days are one of several organ failure-free outcome measures to quantify the efficacy of therapies and interventions. VFDs are typically defined as follows:
  * VFDs = 0 if subject dies within 28 days of mechanical ventilation.
  * VFDs = 28 - x if successfully liberated from ventilation x days after initiation.
  * VFDs = 0 if the subject is mechanically ventilated for >28 days.
Intensive Care Unit mortality | Up to 60 days after randomization
  Mortality rate evaluated during Intensive care unit stay
Day-60 mortality | 60 days after randomization
  Mortality rate evaluated 60 days after randomization
Nosocomial pneumonia | Up to 60 days after randomization
  Number of patients with pneumonia diagnosed during intensive care unit stay
Bacteremia | Up to 60 days after randomization
  Number of patients with bacteremia diagnosed during intensive care unit

OTHER OUTCOMES:
Extra corporeal membrane oxygenation (ECMO) | Up to 60days after randomization
  Placement of ECMO during intensive care unit stay
Tracheostomy | Up to 60 days after randomization
  Number of patients who underwent tracheostomy during intensive care unit stay
Prone Position | Up to 60 days after randomization
  Number of Prone position session

CONTACTS AND LOCATIONS:
Overall Officials: Francois STEPHAN, MD, PhD, Principal Investigator — Centre Chirurgical Marie Lannelongue
Locations (1):
- Reanimation adulte. Hopital Marie Lannelongue, Le Plessis-Robinson, France

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol
Time Frame: Beginning 3 months and ending 24 months following article publication
Access Criteria: Researchers who provide a methodologically sound and proposal. Data are available for 24 months and request should be addressed by email